CLINICAL TRIAL: NCT02591056
Title: An Evaluation of the Combined Effect of the Erchonia® Verju™ Laser With the Green PRESS 8 Lymph Drainage System on the Reduction of Body Circumference
Brief Title: Study of the Combined Effect of Low Level Laser Therapy and Manual Lymph Drainage on Reducing Body Circumference
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC_VERJU+GP8_001
Record Dates: First submitted 2015-10-28; First posted 2015-10-29 (Estimated); Results first posted 2016-09-08 (Estimated); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Circumference Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erchonia Verju Laser + Green PRESS 8 (Experimental): All subjects receive 12 combination treatments over 6 weeks (two per week) with the Erchonia® Verju™ Laser and the Green PRESS 8 devices simultaneously.
  Interventions: Device: Erchonia® Verju™ Laser; Device: Green PRESS 8

INTERVENTIONS:
Device: Erchonia® Verju™ Laser — There are 12 procedure administrations with the Erchonia® Verju™ Laser across 6 weeks: 2 procedures per week. For each procedure administration, the Erchonia Verju is applied to the midsection for 30 minutes: 15 minutes to the front and 15 minutes to the back. All subjects receive the active Erchonia Verju Laser treatment for all 12 procedure administrations.
Device: Green PRESS 8 — There are 12 procedure administrations with the Green PRESS 8 across 6 weeks: 2 procedures per week. For each procedure administration, the Green PRESS 8 is applied to the midsection for 30 minutes. All subjects receive the active Green PRESS 8 treatment for all 12 procedure administrations. Each Green PRESS 8 procedure administration occurs right after each procedure administration with the Erchonia Verju Laser.

SUMMARY:
The purpose of this study is to determine whether low level laser light therapy applied using the Erchonia Verju Laser combined with manual lymph drainage applied using the Iskra Medical Green PRESS 8 Lymph Drainage System is effective in reducing the circumference of the waist, hips and upper abdomen.

DETAILED DESCRIPTION:
The American Society of Plastic Surgeons (ASPS) 2011 report states that the market for cosmetic procedures has shown significant growth over the past two years, with 13.8 million cosmetic plastic surgery procedures performed in the United States in 2011, up 5% since 2010. While surgical cosmetic procedures significantly increased from 2010 to 2011, the overall growth in cosmetic procedures is primarily driven by a substantial rise in minimally-invasive procedures that increased 6%, with nearly 12.2 million cosmetic minimally-invasive procedures having been performed in 2011. This highlights the growing consumer demand for non- or minimally-invasive cosmetic procedures that do not involve surgical procedures such as liposuction and the associated risks, potential complications and lengthy and painful recovery processes.

Low level laser light therapy (LLLT) offers a simple, non-invasive, safe, effective and side-effect free alternative to achieving body circumference reduction. Erchonia low level lasers, including the Erchonia® Verju™ Laser, have been determined safe and effective by the FDA for application for body circumference reduction indications for multiple body areas.

The Iskra Medical Green PRESS 8 is a manual lymph drainage system that is also a simple, non-invasive, safe and side-effect free alternative to achieving body circumference reduction that has demonstrated optimal effectiveness when used in combination with other established alternative non-invasive means of body circumference reduction such as LLLT application.

LLLT, as applied with the Erchonia® Verju™ Laser, effects a transitory pore in the adipocyte cell membrane that enables the fat to pass from the intracellular space into the extra-cellular space. The Green PRESS 8 operates according to the principle of manual lymph drainage, employing pumping of air under controlled pressure into inflatable cuffs according to pre-set pressure, compression pause duration and therapy time parameters. The alternating release and compression of the different vascular and lymphatic structures effects and enhances lymphatic drainage that results in an influx of blood along with nourishing elements, and the elimination of fluids and metabolic waste products. When used in combination with LLLT, this process enhances and accelerates the process of reduction in the size of adipocyte cells through increased liquefaction and emulsification of the fat through the transitory pore in the adipocyte cell, which has been initiated by the preceding application of LLLT.

The purpose of this study is to evaluate if green diode LLLT as applied with the Erchonia® Verju™ Laser is more effective on reducing the circumference of the hips, waist and upper abdomen when used in combination with the Green PRESS 8 manual lymph drainage system twice weekly for six weeks than when used alone.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 25 kg/m² and 40 kg/m², inclusive.
* Subject indicated for liposuction or use of liposuction techniques for the removal of localized deposits of adipose tissues that do not respond to diet and exercise; specifically for the indication of body contouring in the areas of the hips, waist and upper abdomen. (As per the American Academy of Cosmetic Surgery's 2006 Guidelines for Liposuction Surgery developed by A joint Ad Hoc Committee of the American Society of Lipo-Suction Surgery (ASLSS) and the American Academy of Cosmetic Surgery (AACS))
* Subject is willing and able to abstain from partaking in any treatment other than the study procedures (existing or new) to promote body contouring/circumference reduction/weight loss during the course of study participation.
* Subject is willing and able to maintain his or her regular (typical pre-study) diet and exercise regimen without effecting significant change in either direction during study participation.

Exclusion Criteria:

* Known cardiovascular disease such as cardiac arrhythmias, congestive heart failure.
* Cardiac surgeries such as cardiac bypass, heart transplant surgery, pacemakers.
* Prior surgical intervention for body sculpting/weight loss, such as liposuction, abdominoplasty, stomach stapling, lap band surgery, etc.
* Medical, physical, or other contraindications for body sculpting/weight loss.
* Current use of medication(s) known to affect weight levels/cause bloating or swelling and for which abstinence during the course of study participation is not safe or medically prudent.
* Any medical condition known to affect weight levels and/or to cause bloating or swelling.
* Diagnosis of, and/or taking medication for, irritable bowel syndrome.
* Active infection, open wound (e.g. sores, cuts, ulcers, burns, etc.) or other external trauma to the areas to be treated with the laser/lymphatic drainage system devices.
* Known photosensitivity disorder.
* Current active cancer or currently receiving treatment for cancer.
* History of blood clots or phlebitis, other bleeding disorder
* Pregnant, possibly pregnant or planning pregnancy prior to the end of study participation.
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in past two years.
* Developmental disability or cognitive impairment that in the opinion of the investigator would preclude adequate comprehension of the informed consent form and/or ability to record the necessary study measurements.
* Involvement in litigation and/or a worker's compensation claim and/or receiving disability benefits related to weight-related and/or body shape issues.
* Participation in a clinical study or other type of research in the past 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory C Roche, DO, Principal Investigator
Locations (3):
- United States (3):
  - Stockton Plastic Surgery, Stockton, California
  - Cosmetic Surgery, Marion, Indiana
  - Bloomfield Laser and Cosmetic Surgery Center, Bloomfield Hills, Michigan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Erchonia Verju Laser + Green PRESS 8: All subjects receive 12 combination treatments over 6 weeks (two per week) with the Erchonia® Verju™ Laser and the Green PRESS 8 devices simultaneously.
  Erchonia Verju Laser + Green PRESS 8: There are 12 combined procedure administrations with the Erchonia® Verju™ Laser and the Green PRESS 8 simultaneously across 6 weeks: 2 procedures per week. For each procedure administration, the Erchonia Verju is applied to the midsection for 30 minutes: 15 minutes front and 15 minutes back, followed by administration of the Green PRESS 8 to the midsection for 30 minutes. All subjects receive the combination Erchonia Verju Laser + Green PRESS 8 treatment for all 12 procedure administrations.
Period: Overall Study
Arm/Group | Erchonia Verju Laser + Green PRESS 8
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erchonia Verju Laser + Green PRESS 8
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.15 (13.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27
Combined Circumference [Mean (Standard Deviation); unit: inches] — Measurements in inches were taken for the subject's waist, hips and upper abdomen and added together to get a combined circumference measurement.
  inches | 112.34 (13.67)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.64 (3.97)

OUTCOME MEASURES:

1. Primary Outcome: Change in Combined Circumference Measurements
Description: Combined circumference measurement is calculated as the sum of the measurements for the individual body areas of the hips, waist and upper abdomen. Change in combined circumference measurements is calculated as the difference in measurements from baseline to after completion of the 6-week procedure administration period. A negative (-) change indicates a reduction in combined circumference measurement across the evaluation period and is positive for study success. A positive (+) change indicates an increase in combined circumference measurements across the evaluation period and is negative for study success. A mean change for the study subject group of -3.0 inches or more in combined circumference measurements will be considered a clinically meaningful and statistically significant positive change indicative of study success.
Time Frame: Baseline and 6 Weeks
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Erchonia Verju Laser + Green PRESS 8
Number analyzed (Participants) | 27
inches | -3.88 (2.70)
Statistical Analysis 1: Comparison: Erchonia Verju Laser + Green PRESS 8; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; t=+7.45; df=26

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Erchonia Verju Laser + Green PRESS 8
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No